CLINICAL TRIAL: NCT03930342
Title: Native-Changing High-risk Alcohol Use and Increasing Contraception Effectiveness Study
Acronym: Native-CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: University of Colorado, Denver (Other); Sanford Research (Other); Missouri Breaks Industries Research, Inc. (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Michael McDonell, Principal Investigator, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17162-001
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Contraceptive Usage; Alcohol Use Complicating Childbirth; Alcohol Drinking
MeSH Terms: conditions — Contraception Behavior; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Women will be randomized 1:1 to the intervention or usual care conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Native CHOICES Intervention (Experimental): Native-CHOICES will comprise usual care plus 2 MI sessions delivered over 4 weeks; a contraception counseling session at a local clinic; and 3 months of electronic messaging to boost the effects of MI and counseling by increasing perceptions of social connection and social support for behavior change. Contraception counseling will be completed within 2 weeks after the second MI session, so the maximum duration of MI and counseling for each participant will be 6 weeks. Electronic messaging will include positive motivational content consistent with alcohol and contraception use goals set in the MI sessions.
  Interventions: Behavioral: Native-CHOICES
- Wait-list Control Group (No Intervention): The control condition will comprise usual care for the 6-month study period, with a wait-list design that offers women the Native- CHOICES program after they have completed the 6-month data collection.

INTERVENTIONS:
Behavioral: Native-CHOICES — Native CHOICES is a behavioral intervention for prevention of prenatal alcohol exposure in women at high risk for alcohol-exposed pregnancies. The intervention uses motivational interviewing and cognitive-behavioral strategies, and targets adoption of effective contraception and reduction of alcohol use.
  Arms: Native CHOICES Intervention

SUMMARY:
Native CHOICES is a randomized controlled trial of an adapted intervention to reduce the risk of alcohol exposed pregnancies in American Indians and Alaska Natives (AI/ANs). We will enroll 350 AI/AN women living on the Cheyenne River Sioux Indian Reservation or in Rapid City in South Dakota who are 18-44 years old, have risky drinking behaviors, are not currently pregnant but are able to become pregnant, and are sexually active but not using effective contraception.

DETAILED DESCRIPTION:
Fetal alcohol spectrum disorder (FASD) prevalence is up to 10 times higher in American Indians and Alaska Natives (AI/ANs) than in the general US population, yet FASD is 100% preventable. Even moderate alcohol use during pregnancy can affect fetal growth and behavioral outcomes. Alcohol use disorders and binge drinking in women are among the strongest risk factors for FASD in their offspring. AI/ANs have the highest prevalence of alcohol use disorders among US racial and ethnic groups, and are the most likely to engage in binge drinking during pregnancy. A growing consensus indicates that prevention of alcohol-exposed pregnancy must begin before conception. One promising approach is the Changing High-risk Alcohol Use and Increasing Contraception Effectiveness Study (CHOICES), which combines motivational interviewing with contraception counseling for non-pregnant women. In a randomized trial, women receiving CHOICES were 36% more likely to have reduced risk for alcohol-exposed pregnancies after 6 months than women receiving usual care, but the trial did not enroll AI/ANs or rural women. Although the Centers for Disease Control and Prevention has recommended its dissemination, the public health value and cost-effectiveness of CHOICES in AI/ANs is unknown. We propose a randomized controlled trial of an adapted intervention - Native-CHOICES - to reduce risk of alcohol exposed pregnancies in AI/ANs. We will enroll 350 AI/AN women living on the Cheyenne River Sioux Indian Reservation or in Rapid City in South Dakota who are 18-44 years old, have risky drinking behaviors, are not currently pregnant but are able to become pregnant, and are sexually active but not using effective contraception. Native-CHOICES will consist of 2 motivational interviewing sessions plus 1 contraceptive counseling session over 4 weeks, with supportive electronic messaging for 3 months to increase perceived social connectedness and support for modifying drinking behavior and using contraception.

ELIGIBILITY:
Inclusion Criteria:

* Native American Woman
* 18-44 years old at the time of recruitment
* Self-report high-risk drinking behavior (average 8 or more drinks per week) or episodes of binge drinking (four or more drinks on a single occasion) in the past 90 days
* Have vaginal sex with a male partner in the past 30 days

Exclusion Criteria:

* Diagnosed as infertile
* Pregnant
* Effectively using contraceptives defined by standard methods
* Living in a household with someone who is already enrolled in the study

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 404 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonell, MD, Principal Investigator — Washington State University
Locations (2):
- United States (2):
  - Missouri Breaks Industries Research Inc, Eagle Butte, South Dakota
  - Missouri Breaks Industries Research Inc, Rapid City, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Native CHOICES Intervention: Native-CHOICES will comprise usual care plus 2 Motivational Interviewing (MI) sessions delivered over 4 weeks; a contraception counseling session at a local clinic; and 3 months of electronic messaging to boost the effects of MI and counseling by increasing perceptions of social connection and social support for behavior change. Contraception counseling will be completed within 2 weeks after the second MI session, so the maximum duration of MI and counseling for each participant will be 6 weeks. Electronic messaging will include positive motivational content consistent with alcohol and contraception use goals set in the MI sessions.
  Native-CHOICES: Native CHOICES is a behavioral intervention for prevention of prenatal alcohol exposure in women at high risk for alcohol-exposed pregnancies. The intervention uses motivational interviewing and cognitive-behavioral strategies, and targets adoption of effective contraception and reduction of alcohol use.
Period: Overall Study
Arm/Group | Native CHOICES Intervention | Wait-list Control Group
Started | 205 | 199
Three Month Follow-up | 155 | 139
Six Month Follow-up | 150 | 139
Completed (Completed here means participants who completed the baseline, 3 month, and 6 month data collection sessions) | 135 | 122
Not Completed | 70 | 77
Not completed — Lost to Follow-up | 70 | 77

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Native CHOICES Intervention | Wait-list Control Group | Total
Number analyzed (Participants) | 205 | 199 | 404
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 205 | 199 | 404
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.6) | 31.8 (6.7) | 31.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 199 | 404
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 19
  Not Hispanic or Latino | 197 | 188 | 385
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 202 | 192 | 394
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 0 | 0 | 0
Risk for Alcohol Exposed Pregnancy [Count of Participants; unit: Participants] — Baseline enrollment criteria required participants to be at risk for an Alcohol Exposed Pregnancy (AEP) via risky drinking behaviors and engaging in sexual activity without effective and consistent contraceptive measures in the past 3 months.
  Participants | 205 | 199 | 404

OUTCOME MEASURES:

1. Primary Outcome: Risk of Alcohol Exposed Pregnancy
Description: Our primary outcome is measurement of change in risk of alcohol exposed pregnancy (AEP). Being at risk for an AEP is defined as engaging in heavy/binge drinking and ineffective contraception use in the 3 months prior to the final data collection session after exposure to the intervention. Count reflects number of participants who remained at risk for an AEP.
Time Frame: Baseline, 3 months and 6 months post intervention
Population: Data was included only for participants who completed both the 3-month and 6-month follow-up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Native CHOICES Intervention | Wait-list Control Group
Number analyzed (Participants) | 135 | 122
Participants | 103 | 99
Statistical Analysis 1: Comparison: Wait-list Control Group; Results here reflect analysis of the relative risk for AEP that is a combination of risk from baseline to the 3 month timepoint and risk between the 3 month timepoint and 6 month timepoint. This reflects changes in AEP risk across the course of exposure to the intervention (baseline to 3 month) and enduring change post-exposure (3 months to 6 months); Test type: Superiority; Regression, Logistic; Used marginal standardization to estimate relative risk from logistic regression; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.83 to 1.07]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected through each participant's 6-month participation in the study.
Description: Adverse events were largely made known through field staff's personal connection to the community.
Arm/Group | Native CHOICES Intervention | Wait-list Control Group
All-Cause Mortality (participants affected / at risk) | 6/207 | 2/201
Serious Adverse Events (participants affected / at risk) | 1/207 | 0/201
Other Adverse Events (participants affected / at risk) | 0/207 | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Native CHOICES Intervention (N=207) | Wait-list Control Group (N=201)
Heart Attack (Cardiac disorders) | 1 (1) | 0 (0) — At a follow up phone call visit the participant informed field staff that they were hospitalized with a heart attack.

LIMITATIONS AND CAVEATS:
The COVID pandemic hit mid-data collection and this meant that the intervention that was planned for exclusively in-person delivery had to be adapted for delivery over the telephone which may have impacted the results.

This study was also regionally and culturally specific to AI communities in the Northern Plains.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2024-12-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03930342/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03930342/SAP_001.pdf
  • Informed Consent Form: In Person Version (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03930342/ICF_002.pdf
  • Informed Consent Form: Remote Version (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT03930342/ICF_003.pdf